CLINICAL TRIAL: NCT00628121
Title: Clinical Pharmacological Study of NS75A for Healthy Adult Women
Brief Title: Clinical Pharmacological Study of GnRH Antagonist, Cetrorelix for Healthy Female Volunteer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Collaborators: Shionogi (Industry); AEterna Zentaris (Industry)
Responsible Party: Nippon Kayaku Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9575A402
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Premenopause
Keywords: infertility, menstrual cycle, LH surge
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cetrorelix 1 mg (Experimental)
  Interventions: Drug: Cetrorelix
- Cetrorelix 2 mg (Experimental)
  Interventions: Drug: Cetrorelix
- Cetrorelix 3 mg (Experimental)
  Interventions: Drug: Cetrorelix

INTERVENTIONS:
Drug: Cetrorelix — 1, 2 or 3mg, subcutaneouly dosed with single dose
  Other Names: NS75A

SUMMARY:
GnRH analogs are globally used for assisted reproduction in infertile patients. To date, in healthy female volunteers the pharmacokinetic and pharmacodynamic profiles of cetrorelix when administered in a single dose have been investigated in studies conducted using doses of 1, 3 and 5 mg. Studies performed in premenopausal female volunteers confirmed that cetrorelix rapidly suppresses luteinizing hormone (LH) and estradiol and shows dose-dependent prolongation of the duration of LH suppression. However, there have been few reports of studies of the relationship between the cetrorelix dosage and its effect on LH surge. In the present study, we investigated the effect of cetrorelix on LH surge when this drug was administered in single doses of 1, 2 and 3 mg.

DETAILED DESCRIPTION:
To evaluate that effect on LH surge, we investigated the efficacy of cetrorelix in delaying the start of the LH surge in comparison with the control menstrual cycle when saline was administered, and also examined the mode of disappearance of pulsatile LH secretion during the cetrorelix administration menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* a BMI of 18 years old and <18 and 25 years old and >25
* menstrual cycles was within the range of 25~31 days

Exclusion Criteria:

* use of a drug (e.g., oral contraceptives, drugs for treatment of hyperprolactinemia, GnRH agonists, sex steroid hormones, psychoactive drugs, etc.)
* serious disease of the endocrine system, liver, kidney, heart, lung, digestive system, etc.
* a generalized drug allergy

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-04; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Day of the LH surge | Saline administration menstrual cycle, cetrorelix administration menstrual cycle

SECONDARY OUTCOMES:
Serum LH concentrations | Saline administration menstrual cycle, cetrorelix administration menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Kitasato University East Hospital, Sagamihara, Kanagawa, Japan